CLINICAL TRIAL: NCT02312570
Title: A Prospective, Randomized Clinical Trial of PRP Concepts Fibrin Bio-Matrix in Chronic Non-Healing Pressure Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PRP Concepts, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC004
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Pressure Ulcer
Keywords: non-healing wounds; pressure ulcer; platelet rich plasma
MeSH Terms: conditions — Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PRP Concepts Fibrin Bio-Matrix (Experimental): PRP Concepts Fibrin Bio-Matrix in addition to usual and customary practice
  Interventions: Device: PRP Concepts Fibrin Bio-Matrix; Other: Usual and Customary Practice
- Usual and Customary Practice (Other): Usual and customary practice for non-healing pressure wounds
  Interventions: Other: Usual and Customary Practice

INTERVENTIONS:
Device: PRP Concepts Fibrin Bio-Matrix — Administration of PRP Concepts Fibrin Bio-Matrix to wound in addition to usual and customary care
  Arms: PRP Concepts Fibrin Bio-Matrix
Other: Usual and Customary Practice — Ussual and customary care of non-healing pressure wounds
  Other Names: Standard of Care

SUMMARY:
To assess the efficacy of the PRP Concepts Fibrin Bio-Matrix and compare its performance with usual and customary practice for the treatment of chronic non-healing pressure ulcers (PU).

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, controlled, multi-center study for subjects undergoing PU treatment. Qualified subjects will be randomized (1:1); test group (PRP Concepts Fibrin Bio-Matrix) and control group (usual and customary practice). The study will consist of 3 periods: a screening period, an active treatment period, and a follow-up period (if healed). Approximately 250 subjects will be enrolled. Subjects will be ≥18 years of age with a PU (greater than 4 weeks duration). Each subject will be enrolled in the active treatment period for up to 12 weeks, or to closure of wound with a confirmatory visit 2 weeks after wound closure, whether such closure occurs at 12 weeks or earlier.

ELIGIBILITY:
Inclusion Criteria:

Medicare/Medicaid eligible Ulcer of pressure/shear etiology The index ulcer is greater than 4 weeks duration. Three or fewer ulcers that are separated by > 3.0 cm distance The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) that is located on the heel, ischium, sacrum, and trochanter Post-debridement, the ulcer size must be between 2 cm2 and 200 cm2 Demonstrated adequate offloading regimen Able and willing to attend scheduled follow-up visits and study related exams Able and willing to provide a voluntary written informed consent

Exclusion Criteria:

Stage I pressure ulcers Ulcers that are unstageable or of deep tissue morphology that have yet to become an open wound Ulcer not of PU pathophysiology (e.g., pure diabetic, vasculitic, radiation, rheumatoid, collagen vascular disease, venous, or arterial etiology) Greater than 30% reduction in wound size during the first two weeks of observation and treatment by the investigator Gross clinical infection at the study ulcer site including cellulitis and osteomyelitis. Known allergy tor sensitivity to Eclipse PRP kit components (calcium chloride, calcium gluconate or acid citrate dextrose solution A (ACDA)) Serum albumin of less than 2.5 g/dL, Plasma Platelet count of less than 100 x 109/L, Hemoglobin of less than 10.5 g/dL Known renal failure as determined by a Creatinine > 2.5 mg/dl Malignancy at or near the ulcer site Rheumatoid arthritis (and other collagen vascular disease), vasculitis, sickle cell disease, HIV Severe liver disease. Presence of additional abnormal lab values obtained within 7 days prior to the Day 0 visit determined to be clinically significant by the investigator including: WBC >13,000/cm3 or < 5, 000 cm3, or electrolytes that are outside the host institution's range of normal Radiation therapy, chemotherapy, immunosuppressive therapy or chronic steroid use within 30 days of enrollment Received another investigational device or drug within 30 days of enrollment Received allograft, autograft or xenograft within 30 days of enrollment Subject has inadequate venous access for repeated blood draw required for Eclipse RPR administrations Subject requires or is anticipated to require interventions directed at improvement of arterial perfusion to affected area Ulcer expected to be treated with any advanced therapeutics (e.g., HBOT) Presence of another wound that is concurrently treated and might interfere with treatment of index wound Subjects who are cognitively impaired and do not have a healthcare proxy Life expectancy of < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent of wounds that have healed at 12 weeks | 12 weeks
  To assess the efficacy and safety of an autologous PRP membrane matrix treatment by measurement and observation of time to and percent of complete wound closure, wound healing trajectory, and wound recurrence over time as compared to the standard of care non-healing wound treatment.
To assess by a validated interview-scoring tool, the changes in quality of life and ability to return to previous function/resumption of normal activities. | 12 weeks
  To assess by a validated interview-scoring tool, the changes in quality of life and ability to return to previous function/resumption of normal activities

SECONDARY OUTCOMES:
Wound trajectory (Mean Change) | 12 weeks
  Mean of percent (%) wound size changes at 4 weeks, 8 weeks and 12 weeks
Wound trajectory (Median Change) | 12 weeks
  Median of percent (%) wound size changes at 4 weeks, 8 weeks and 12 weeks
Ulcer recurrence | 3 months
  Ulcer recurrence out to 3 months for subjects whose wounds heal by conclusion of 12 week visit.
Quality of Life Health Survey | 3 months
  Changes in Quality of Life scores and ability to return to previous function/resumption of normal activities

CONTACTS AND LOCATIONS:
Overall Officials: Damon Keeley, Study Director — PRP Concepts, LLC
Locations (1):
- Westchester General Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No